CLINICAL TRIAL: NCT00509132
Title: A Phase I, Double-Blind, Randomized, Placebo-Controlled Ascending IV Single-Dose Tolerance and Pharmacokinetic Study of Trodusquemine in Healthy Volunteers
Brief Title: A Tolerance and Pharmacokinetic Study of Trodusquemine in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genaera Corporation (Industry)
Responsible Party: Michael Gast, MD, PhD, Genaera Corporation
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MSI-1436C-101
Record Dates: First submitted 2007-07-27; First posted 2007-07-31 (Estimated); Last update posted 2008-01-09 (Estimated); Status verified 2008-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — 3-N-1(spermine)-7, 24-dihydroxy-5-cholestane 24-sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: trodusquemine

SUMMARY:
The purpose of this study is to evaluate the safety and tolerance of single intravenous (through a vein) doses of trodusquemine. Different amounts of trodusquemine will be given to each volunteer group throughout the study. Another purpose is to evaluate the pharmacokinetics (PK - the study of the way the drug enters and leaves the blood and tissues over time) of trodusquemine. Finally, this study will also determine whether trodusquemine has any effect on appetite, mood or behavior, and selective biomarkers (substances in your blood that may change in response to the study drug).

ELIGIBILITY:
Inclusion Criteria:

* male or female subjects, between 18 and 55 years old (inclusive);
* body mass index (BMI) of 27-40 kg/m2;

Exclusion Criteria:

* likely allergy or sensitivity to any components of Trodusquemine for Injection based on known allergies to drugs of the same class, or which, in the opinion of the Principal Investigator, suggests an increased potential for an adverse hypersensitivity to trodusquemine HCl;
* any subject with a history of allergy (rash, hives, breathing difficulty, etc.) to any medications, either prescription or nonprescription, including dietary supplements or herbal medications;
* any subject with a history of severe allergy or bronchial asthma;

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2007-05; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phil Leese, MD, Principal Investigator — Quintiles, Inc.
Locations (1):
- Quintiles, Inc., Overland Park, Kansas, United States